CLINICAL TRIAL: NCT00511732
Title: A Randomized, Double-blind, Controlled, Stepwise Titration Study to Evaluate Dose Response to Prandial Administration of Inhaled Technosphere/Insulin or Technosphere in Patients With Type 2 Diabetes Mellitus Who Are Sub-optimally Treated
Brief Title: 18-Week, Randomized, Double-blind, Placebo Controlled, Forced Titration Study of Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MKC-TI-005
Record Dates: First submitted 2007-08-03; First posted 2007-08-06 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Technosphere Insulin (Experimental)
  Interventions: Drug: Technosphere Insulin
- Technosphere Inhalation Powder (Placebo Comparator)
  Interventions: Drug: Technosphere Placebo

INTERVENTIONS:
Drug: Technosphere Insulin — Technosphere Insulin Inhalation Powder
  Arms: Technosphere Insulin
Drug: Technosphere Placebo — Technosphere Inhalation Powder
  Arms: Technosphere Inhalation Powder

SUMMARY:
Designed to evaluate dose response of force-titrated prandial administration of TI as compared to placebo (TP) in subjects with Type 2 diabetes who were suboptimally controlled

ELIGIBILITY:
Inclusion Criteria:

* Male and females patients from 18 to <80 years of age
* Clinical diagnosis of type 2 diabetes mellitus
* Duration of diabetes of >3 years and <20 years
* Glycemic control at upper end of acceptable level or sub-optimal in control (HbA1c between 7.0% and 12?0%)
* Confirmation of diagnosis of diabetes such as a history of 2 hour postprandial blood glucose >11.1 mmol/L (200 mg/dL) or following a glucose tolerance test
* A minimum of 2 months of treatment with a stable dose of one or more of the following anti-hyperglycemic agents: sulphonylureas, alpha glucosidase inhibitors, metformin, meglitinides, thiazolidinediones and/or Lantus basal insulin therapy
* FBG:>6 mmol/L (108 mg/dL)
* C-peptide: >0.5 nmol/L
* BMI <38 kg/m2
* Baseline DLco, FVC, FEV1 >75% of predicted normal
* Subjects who, in the opinion of the Investigator, will be able to complete this study
* Written informed consent

Exclusion Criteria:

* Severe complications of diabetes including history of: blindness from or grade III or IV diabetic retinopathy, renal failure requiring dialysis or transplantation, amputation of limbs or digits related to diabetic vasculopathy or foot ulcers
* Treatment with another investigational drug within 3 months prior to study entry and for the duration of the study
* History of drug or alcohol dependency
* Significant hepatic disease (as evidenced by ALT or AST >3 times the normal upper reference range or bilirubin >1.5 times the normal upper reference range)
* Significant renal disease (as evidenced by creatinine >1.5 mg/dL for males or >1.3 mg/dL for females) or proteinuria >1,000 mg/24 hours
* History of chronic obstructive pulmonary disease, or history of other known chronic pulmonary diseases, such as reactive airway disease, chronic bronchitis, emphysema, or asthma
* Heart disease graded as class III or class IV according to New York Heart Association criteria
* Prior treatment with , or participation in a clinical study involving an inhaled insulin product
* Smokers
* Current use of preprandial or prandially administered fast-acting or rapid acting insulin or insulin analogs
* Previous participation in a TI or TP clinical trial
* Allergy to insulin or to any drugs to be used as part of the clinical trial
* History of malignancy within 5 years of study entry (other than basal cell carcinoma)
* Anemia (hemoglobin level less than 11 g/dL for females or 12 g/dL for males at study entry)
* Diagnosis of Acquired Immunodeficiency Syndrome (AIDS) and Aids Related Complex A major psychiatric disorder that will preclude satisfactory participation in this study
* Subjects who have had a myocardial infarction or stroke within the preceding 6 months
* Prior diagnosis of systemic autoimmune or collagen vascular disease requiring previous or current treatment with systemic corticosteroids, cytotoxic drugs, or penicillamine
* History of severe or multiple allergies
* Progressive fatal disease
* Recent loss (within the past 2 months) of >5% of body weight
* Evidence of "moderate" or greater ketones in urine or history of ketoacidosis
* Use of medications known to modify glucose metabolism or the ability to recover from hypoglycemia such as oral, parenteral and inhaled steroids, or greater than 25 mg hydrochlorothiazide daily
* Women who are pregnant or lactating
* Women of childbearing potential practicing inadequate birth control (adequate birth control is defined as using oral contraceptives, condoms or diaphragms with spermicide, intrauterine devices, or surgical sterilization).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2004-06; Primary Completion 2005-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
HbA1c change from baseline (week 6) to end of treatment (week 17) | measured from week 6 (baseline) to week 17
Area under the plasma glucose concentration versus time (AUCglucose) compared to week 6 (baseline. | at weeks 4, 6, 11 and 17
  Timepoints: 0 minutes (before meal) and at 15, 30, 60, 90, 120, 180, 240, and 300 minutes after TI administration
Area under the plasma glucose concentration versus time (AUCglucose) compared to week 6 (baseline) | at weeks 4, 6, 11 and 17
  Timepoints: 0 minutes (before meal) and at 15, 30, 60, 90, 120, 180, 240, and 300 minutes after Technosphere Placebo administration

SECONDARY OUTCOMES:
Fasting blood glucose concentration compared to week 6 (baseline) | at weeks 4, 6, 11 and 17
Safety variables included adverse events (AEs), clinical laboratory tests, vital signs and physical examinations | 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anders Boss, Study Director — Mannkind Corporation